CLINICAL TRIAL: NCT05574790
Title: Identification of Multimorbid Patients With a Higher Probability of Readmission and Mortality: Role of Patient-related Variables
Brief Title: Identification of Multimorbid Patients With a Higher Probability of Readmission and Mortality
Status: Completed | Type: Observational
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Collaborators: Hospital Costa del Sol (Other); Hospital del Mar (Other); Instituto de Salud Carlos III (Other Government); Hospitales Universitarios Virgen del Rocío (Other); Asociacion Instituto de Investigacion en Servicios de Salud Kronikgune (Unknown)
Responsible Party: Principal Investigator, Susana García Gutiérrez, principal investigator, Hospital Galdakao-Usansolo
Other Study IDs: PI18/01438
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Multimorbidity
Keywords: multimorbid Patients; Readmission; Mortality; Predictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Admitted: We will include patients who had been admitted by meeting Ollero et al categories in hospitalization ward
  Interventions: Other: annual follow up

INTERVENTIONS:
Other: annual follow up — Collection of the following information during the year following discharge from the initial episode (initial cohort): readmissions, dates and causes of readmission, mortality

SUMMARY:
A prospective qualitative quantitative study was designed to create predictive models of readmission in multimorbid patients.

DETAILED DESCRIPTION:
Social determinants have been shown to be related to the probability of readmission and death in multimorbid patients. These are increasingly older, which makes them more likely to be readmitted when their preferences are usually to be at home. Objective: To create and validate prediction models for readmission and mortality during home transitional period (1 month) and up to a year, in multimorbid patients, including variables related to the patient and their social environment. Design: Quali-quantitative. 4 hospitals from 3 regions (Andalucia, Catalonia and the Basque Country) will participate . Patients presenting at least 2 of the Ollero's categories will be included. Variables will be identified by means of nominal groups of professionals and focal groups with patients and caregivers. These variables will be included in the final models join to clinical variables, PROMS (health related quality of life, burden of the caregiver , social support). Logistic/ Cox regression models will be developed and validated internally to identify the risk of readmission and death which will be validated in an external cohort. Expected results: We hope to provide the health system with stratification tools for polypathological patients that help in identifying those patients with the greatest need for individualized interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients discharged from the Internal Medicine departments of the participating centers due to acute pathology, de novo or decompensation of a chronic pathology who also present at least 2 of the cathegories of Ollero et al.

Exclusion Criteria:

* Patients admitted for end-of-life treatment, scheduled admissions, exacerbation of rheumatic pathology or systemic disease, study of anaemia in patients with no-known comorbidity, search for neoplasia and acute processes without associated comorbidity. -
* Failure to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: multimorbid patients who are equivalently complex and with high risk for destabilization, difficult to manage and with mutual interrelationships.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Readmission | 1 month
  number of readmissions in the early period (transition to discharge, 1 month
Readmission | 1 year
  number of readmissions in the annual period

CONTACTS AND LOCATIONS:
Overall Officials: Susana García Gutiérrez, PhD, Principal Investigator — Unidad de Investigación. Hospital Galdakao-Usansolo. Osakidetza
Locations (4):
- Spain (4):
  - Hospital Galdakao Usansolo, Galdakao, Bizkaia
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital del Mar, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: Undecided